CLINICAL TRIAL: NCT03002064
Title: Docetaxel Plus Cisplatin Versus 5-fluorouracil Plus Cisplatin as First-line Treatment for Metastatic Esophageal Squamous Patients: a Prospective Multicenter, Randomized Controlled Clinical Study
Brief Title: Docetaxol Plus Cisplatin Versus 5-Fu Plus Cisplatin as 1st-line Chemotherapy in Advanced ESCC Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ruihua Xu, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-ESO-01
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Esophagus Cancer; Chemotherapy Effects
Keywords: Esophagus squamous carcinoma; First-line chemotherapy; Docetaxel; Cisplatin; 5-fluorouracil
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Docetaxel; Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- DP group (Experimental): Docetaxel plus cisplatin. Docetaxel: 60mg per square metre on day 1 and Cisplatin: 60mg per square metre on day 1, repeated every 3 weeks till progression or at most 6 cycles.
  Interventions: Drug: Docetaxel; Drug: Cisplatin
- PF group (Active Comparator): Cisplatin plus 5-fluorouracil. Cisplatin: 60mg per square metre on day 1 and 5-fluorouracil 3750mg per square metre, civ 120 hours every 3 weeks till progression or at most 6 cycles.
  Interventions: Drug: Fluorouracil; Drug: Cisplatin

INTERVENTIONS:
Drug: Docetaxel — 60mg per square metre on day 1, repeated every 3 weeks till progression or at most 6 cycles.
  Other Names: Docetaxol
  Arms: DP group
Drug: Fluorouracil — 5-fluorouracil 3750mg per square metre, civ 120 hours every 3 weeks till progression or at most 6 cycles
  Other Names: 5-Fu
  Arms: PF group
Drug: Cisplatin — Cisplatin: 60mg per square metre on day 1, repeated every 3 weeks till progression or at most 6 cycles
  Other Names: DDP

SUMMARY:
This is a phase III clinical trial to compare the efficacy of docetaxel plus cisplatin versus 5-Fu plus cisplatin in the first line chemotherapy for advanced or metastatic esophageal squamous carcinoma patients.

DETAILED DESCRIPTION:
Esophageal cancer is the 6th most common cause of cancer deaths worldwide and it is an endemic in many parts of the world, particularly in the developing countries, including China. Histologically, esophageal cancer can be classified as adenocarcinoma and esophageal squamous cell. carcinoma (ESCC) which is the most common histology in Asia. For locally advanced or metastatic ESCC patients, chemotherapy can improve overall survival (OS) and progression free survival (PFS). There is no standard first-line chemotherapy for ESCC patients. Cisplatin (DDP) plus fluorouracil is the most common used combination with a response rate of 25-35%. Previous studies showed that the combination of paclitaxel with cisplatin had good tolerance and efficacy to esophageal carcinoma. This is a prospective randomized control phase III clinical trial to compare the efficacy and safety between docetaxel/cisplatin and 5-Fu/cisplatin as the 1st line treatment in advanced or metastatic esophageal carcinoma patients.

Sample size:

This is a non-inferior study. The planned sample size was 358 patients, allowing for a 10% dropout rate and assuming the median progression free survival was 5.5 months in the experimental group and 4 months in the control group with a hazard ratio of 0.727, α=0.05, β=0.2. The planned enrolled time was 36 months and 12 months of follow up. The ratio between control and experimental group is 1:1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give written informed consent signed voluntarily by patients themselves or their supervisors witted by doctors.
2. Patients must have histologically confirmed esophageal squamous cell carcinoma without prior treatments including surgery, chemotherapy, radiotherapy, and targeting treatment. Patients were allowed to have palliative radiotherapy 3 months before the enrollment and the target lesions should not be within the radiotherapy region. The last date of adjuvant therapy should be over 6 months before the enrollment.
3. With measurable or evaluable disease according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
4. With an expected life expectancy of ≥ 3 months.
5. With a performance status of 0-1 on the Eastern Cooperative Oncology Group (ECOG) scale.
6. Without serious system dysfunction and could tolerate chemotherapy.
7. Patients must have normal bone marrow function with a hemoglobin (HGB) of ≥90g/L, an white blood cell (WBC) counts of ≥4.0×10^9/L，a neutrophil count of ≥2.0×10^9/L, , a platelet count of ≥100×10^9/L.
8. Patients must have normal liver and renal function with a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL), a creatinine (Cr) of ≤ 1.0 UNL, alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤2.5 UNL.
9. Patients must have normal electrocardiogram results and no history of congestive heart failure.
10. Women of childbearing age should voluntarily take contraceptive measures. Without drug addition
11. Patients must be with good compliance and agree to accept follow-up of disease progression and adverse events.

Exclusion Criteria:

1. Allergic to known drug
2. Patients who have received prior treatment including chemotherapy, radiotherapy and surgery for the advanced or metastatic diseases.
3. Receive docetaxel within 6 months as adjuvant or neoadjuvant chemotherapy.
4. Brain metastasis.
5. Without measurable or evaluable disease.
6. With history of other tumors except for those of cervical carcinoma in situ or skin basal cell carcinoma who had been completely treated and without relapse in last 5 years.
7. With serious diseases such as congestive heart failure, uncontrolled myocardial infarction and arrhythmia, liver failure and renal failure.
8. With neurological or psychiatric abnormalities that affect cognitive.
9. Pregnant or lactated women (premenopausal women must give urine pregnancy test before enrollment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 36 months
  From the date of randomization until the date of first documented relapse of disease or date of death from any cause, whichever came first

SECONDARY OUTCOMES:
Overall survival | 36 months
  From the date of randomization until the date of death from any cause.
Response rate | 36 months
  Including complete response and partial response
Grade 3 and 4 toxicities | 36 months
  According to the CTCAE
Quality of life--Score of the questionnaire | 36 months
  EORTC QLQ-C30 and QLQ-OES18 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Rui-Hua Xu, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Cancer center of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No